CLINICAL TRIAL: NCT06128629
Title: MAGNITUDE: A Phase 3, Multinational, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of NTLA-2001 in Participants With Transthyretin Amyloidosis With Cardiomyopathy (ATTR-CM)
Brief Title: MAGNITUDE: A Phase 3 Study of NTLA-2001 in Participants With Transthyretin Amyloidosis With Cardiomyopathy (ATTR-CM)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intellia Therapeutics (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITL-2001-CL-301
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Transthyretin Amyloidosis (ATTR) With Cardiomyopathy
Keywords: TTR; Amyloidosis; Cardiomyopathy; NTLA-2001; ATTR-CM; Transthyretin; ATTR; TTR-mediated amyloidosis; Amyloidosis, Hereditary; Amyloidosis, Hereditary, Transthyretin-Related Amyloidosis; Transthyretin amyloid cardiomyopathy; TTR cardiomyopathy; Wild-type TTR; V122I; Amyloidosis, Wild Type
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis; Cardiomyopathies; Amyloidosis, Familial | interventions — NTLA-2001

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to NTLA-2001 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NTLA-2001 (Experimental): Single intravenous (IV) infusion of NTLA-2001
  Interventions: Biological: NTLA-2001
- Placebo (Placebo Comparator): Single IV infusion of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: NTLA-2001 — NTLA-2001 (55mg) by IV infusion
  Arms: NTLA-2001
Drug: Placebo — Normal saline (0.9% NaCl) by IV infusion
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of a single dose of NTLA-2001 compared to placebo in participants with ATTR-CM.

DETAILED DESCRIPTION:
This is a multinational, multicenter, double-blind, placebo-controlled study in approximately 1200 participants, who will be randomized to receive a single infusion of either NTLA-2001 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of ATTR amyloidosis with cardiomyopathy
* Medical history of heart failure (HF)
* Symptoms of HF are optimally managed and clinically stable within 28 days prior to administration of study intervention
* Screening NT-proBNP, a blood marker of HF severity, greater than or equal to 600 pg/mL and less than 10,000 pg/mL

Exclusion Criteria:

* New York Heart Association (NYHA) Class IV HF
* Polyneuropathy Disability score of IV (confined to wheelchair or bed)
* Has hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* History of active malignancy within 3 years prior to screening
* RNA silencer therapy (patisiran, inotersen and/or eplontersen) within 12 months prior to dosing. Any prior vutrisiran use is not allowed
* Initiation of tafamidis or acoramidis within 56 days prior to study dosing
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2
* Liver failure
* Uncontrolled blood pressure
* Unable or unwilling to take vitamin A supplementation for the duration of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of cardiovascular (CV) mortality and CV events | Maximum study duration is dependent on event rates and is estimated to be at least 18 months and up to 48 months

SECONDARY OUTCOMES:
Change in baseline to month 18 in serum TTR | Baseline, Month 18
Change from baseline to month 18 in KCCQ-OS score | Baseline, Month 18

CONTACTS AND LOCATIONS:
Locations (126):
- United States (37):
  - University of Arizona, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Western Greater Los Angeles VA Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Diego (UCSD) - Medical Center, San Diego, California
  - University of Colorado Denver, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Washington Hospital Center - MedStar Heart and Vascular Institute, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cleveland Clinic of Florida, Weston, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Kentucky Gill Heart Institute, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - New York University (NYU) School of Medicine - Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Oregon Health and Science University (OHSU), Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott and White - The Heart Hospital Baylor Plano, Plano, Texas
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University - Department of Internal Medicine, Richmond, Virginia
- Argentina (6):
  - Fundacion Favalro, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - ICBA, Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma de Buenos Aire
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire
  - Hospital Privado de Rosario, Rosario
- Australia (7):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Westmead Hospital, Westmead, New South Wales
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - The Alfred Hospital, Melbourne
  - Princess Alexandra Hospital, Woolloongabba
- Austria (2):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Universitaesklinikum St. Poelten, Sankt Pölten
- Belgium (5):
  - AZ Sint-Jan Brugge, Bruges
  - Universite Libre de Bruxelles (ULB) - Hopital Erasme, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
- Brazil (9):
  - Centro de Pesquisa NUPEC - Instituto Orizonti em Belo Horizonte, Belo Horizonte
  - Complexo Hospitalar de Niterói (CHN-DASA), Niterói
  - CAPED - Centro Avancado de Pesquisa, Ribeirão Preto
  - HCFMRP - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto, Ribeirão Preto
  - Cardiopulmonar da Bahia S. A. (Hospital Cardio Pulmonar), Salvador
  - Hospital Israelita Albert Einstein, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto do Coracao (InCor) do Hospital das Clinicas da FMUSP, São Paulo
  - PSEG Centro de Pesquisa Clinica S.A., São Paulo
- Canada (4):
  - Alberta Health Services - University of Calgary, Calgary, Alberta
  - Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Fakultni nemocnice u sv. Anny v Brne, Brno, Czechia
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (5):
  - AP-HP Hopital Henri Mondor, Créteil
  - AP-HM - Hopital de la Timone, Marseille
  - AP-HP Hopital Bichat - Claude Bernard, Paris
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - CHU de Toulouse - Hopital Rangueil, Toulouse
- Germany (4):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Semmelweis Egyetem Belgyogyaszati es Hematologiai Klinika, Budapest, Hungary
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital, Ein Karem, Jerusalem
  - Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - Azienda Ospedaliero-Universitaria di Ferrara-Arcispedale Sant'Anna, Cona
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio per la Ricerca Medica, Pisa
  - Azienda sanitaria universitaria Giuliano Isontina (ASU GI) - Ospedale di Cattinara, Trieste
- Japan (4):
  - Kumamoto University Hospital, Kumamoto
  - National Cerebral and Cardiovascular Center, Osaka
  - The University of Tokyo Hospital, Tokyo
  - Toyama University Hospital, Toyama
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico
- Netherlands (3):
  - University Medical Center, Groningen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- New Zealand (2):
  - New Zealand Clinical Research, Auckland
  - New Zealand Clinical Research, Christchurch
- Oslo University Hospital - Rikshospitalet, Oslo, Norway
- Portugal (2):
  - Centro Hospitalar Universitario de Lisboa Norte, Lisbon
  - Centro Hospitalar Universitario do Porto, Porto
- Singapore (2):
  - National Heart Centre, Singapore
  - National University Hospital, Singapore
- Spain (6):
  - Hospital Universitario de A Coruna, A Coruña
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Son Llatzer, Palma de Mallorca
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - University Hospital of Umea, Umeå
- Taiwan (3):
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipai Veterans General Hospital, Taipei
- United Kingdom (7):
  - Synexus Midlands Clinical Research Centre, Birmingham
  - Synexus Wales Clinical Research Centre, Cardiff
  - Synexus Scotland Clinical Research Centre, Glasgow
  - Synexus Hexham Clinical Research Centre, Hexham
  - Synexus Merseyside Clinical Research Centre, Liverpool
  - Richmond Pharmacology, London
  - Synexus Manchester Clinical Research Centre, Manchester

IPD SHARING:
Plan to Share IPD: No